CLINICAL TRIAL: NCT07073144
Title: The Impact of 'Digital Strolling' on Depression and Quality of Life of People With Severe Mobility Impairment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20240930009
Record Dates: First submitted 2025-06-05; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-05

CONDITIONS: Severe Mobility Impairment; Spinal Cord Injuries (Complete and Incomplete); Poliomyelitis
Keywords: severe mobility impairment; virtual reality; depression; quality of life
MeSH Terms: conditions — Spinal Cord Injuries; Poliomyelitis; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual walking group (Experimental): Participants in the virtual walking group will use arm swing locomotion to experience virtual walking in 10 "Digital Strolling" scenarios, mainly in a variety of natural environments.
  Interventions: Behavioral: Virtual walking
- Passive observing group (Active Comparator): Participants in the passive observing group will look at 10 different walking videos.
  Interventions: Behavioral: Passive observing walking

INTERVENTIONS:
Behavioral: Virtual walking — Participants in the intervention group will wear a head-mounted display and hold a controller to swing their arm and control the virtual avatar walking in the virtual world. The intervention will include 10 scenarios of virtual walking intervention (1 scenario daily, each lasting for 15-20 minutes).
  Arms: Virtual walking group
Behavioral: Passive observing walking — Participants in the control group will be given 10 different walking videos in total, one for each day, each approximately 15 minutes in length.
  Arms: Passive observing group

SUMMARY:
This intervention aims to develop and test the feasibility, acceptability, and preliminary effects of a "Digital Strolling" intervention among people with SMI. The intervention group will receive a "Digital Strolling" intervention, which consists of 20 minutes "Digital strolling" for 10 days, with lessons occurring once a day. The control group will receive passive observation of virtual walking videos only.

DETAILED DESCRIPTION:
This study is a two-arm, pilot randomized controlled trial, which will be used to evaluate and compare the effects of the "Digital strolling" intervention and the passive observing control group.

Twenty-four participants will be recruited from the Hong Kong Polytechnic University. Participants will be assigned to the "Digital Strolling" or control group. Participants in the "Digital Strolling" group will receive an arm swing virtual walking intervention, which consists of 20 minutes of virtual walking for 10 days and is conducted at home. Qualitative interviews with the "Digital Strolling" group will be conducted to understand their acceptability, usability, perceived strengths, and limitations of the intervention. While the one in the control group will receive 10 passive observing walking videos for 10 days.

ELIGIBILITY:
Inclusion Criteria:

* Have SMI (people who are inability to walk or climb stairs, stand, or use a wheelchair or scooter by self-report (inability to perform walking or climbing stairs or standing, or use of a wheelchair or scooter) over 6 months
* Have mild to moderate levels of depression
* Able to communicate in Cantonese
* Provide informed consent.

Exclusion Criteria:

* Have severe cognitive impairment
* Have an episode of severe mental illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-05-09 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Depression | Depression will be measured at pre-intervention and 1 week post-intervention.
  Depression will be measured by the 2-item Patient Health Questionnaire and the 9-item Patient Health Questionnaire. The PHQ-2 has two items (depressed mood and anhedonia), with range from 0-6. Highest score represents higher level of depression symptom severity. The PHQ-9 has 9 items (range, 0-27), higher score also means higher level of depression, the severity score ranges are as follows: 0-4 no depression, 5-9 mild depression, 10-14 moderate depression, 15-19 moderately severe depression, and 20-27 severe depression.

SECONDARY OUTCOMES:
Chronic pain | Chronic pain will be assessed at pre-intervention and 1 week post-intervention.
  Chronic pain will be measured using the Numerical Pain Rating Scale (NPRS), with higher score indicate higher pain level, 0 is none pain, 1-3 means mild pain, 4-6 meanes moderate pain, 7-9 means severe pain, 10 is severe and worst pain.
Chronic pain | Chronic pain will be measured at pre-intervention and 1 week post-intervention.
  The chronic pain will also be measured using Brief Pain Inventory (BPI). This scale has two domains: pain severity and pain interference. Mean scores of item 3-6 and 9A-9G reflecting pain severity and pain interference respectively, higher scores indicating higher pain severity or pain interference.
Activity of Daily Living | Activity of Daily Living will be assessed at pre-test and 1 week post-intervention
  Activity of daily living will be measured using the Barthel index, which measures the performance of ten basic activities of daily life (ADL) such as dressing, mobility, and grooming. The total score of this scale ranges from 0-100, 0-20 indicate complete dependence; 21-60 points means severe dependence, 61-90 indicate moderate dependence; 91-99 means mild dependence, 100 points mean complete independence.
Sleep quality | Sleep quality will be assessed at pre-intervention and 1 week post-intervention.
  Sleep quality will be measured using the Pittsburgh Sleep Quality Index. The total score of the scale ranges from 0 to 21; a higher score indicates lower sleep quality.
Quality of life (The 5-level EuroQol of Life -5 dimensions) | Quality of life will be assessed at pre-intervention and 1 week post-intervention.
  Quality of life will be measured using the 5-level EuroQol of Life -5 dimensions. This scale scores ranged from -0.59 to 1, where 1 is the best possible health state.
Anxiety | Anxiety will be assessed pre-intervention and 1 week post intervention
  Anxiety will be measured using the Generalized Anxiety Disorder-7. This scale has 7 items, with a total score ranging from 0-21. 1-4 indicates minimal anxiety, 5-9 indicates mild anxiety, 10-14 indicates moderate anxiety, and 15-21 indicates moderate to severe anxiety.
Virtual presence | Igroup presence questionnaire will be assessed pre-test and 1 week post intervention
  Classifying virtual presence will be assessed using the Igroup presence questionnaire. The questionnaire has three subscales (Spatial presence, involvement, and experienced realism). The questionnaire needs to calculate the average scores across the subscales, then compute an overall sense of presence by averaging these subscale means. Higher subscale means higher spatial presence, involvement, and experienced realism. The higher total scores mean a higher overall sense of presence.
Self-efficacy for exercise | Self-efficacy for exercise scale will be assessed pre-test and 1 week post-intervention
  Self-efficacy for exercise scale will be measured using the Chinese self-efficacy for exercise scale. The total score of this scale ranges from 0 to 90; a higher score represents strong exercise self-efficacy.
Loneliness | Loneliness will be assessed pre-test and 1 week post-intervention
  Loneliness will be measured using the Chinese version of the 6-item De Jong Gierveld Loneliness Scale. This scale has two subscales (emotional loneliness and social loneliness). The scores range from 0 to 6, where 0 means no loneliness and 6 indicates severe loneliness.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Nursing, The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] KATZ S, FORD AB, MOSKOWITZ RW, JACKSON BA, JAFFE MW. STUDIES OF ILLNESS IN THE AGED. THE INDEX OF ADL: A STANDARDIZED MEASURE OF BIOLOGICAL AND PSYCHOSOCIAL FUNCTION. JAMA. 1963 Sep 21;185:914-9. doi: 10.1001/jama.1963.03060120024016. No abstract available. PMID 14044222
- [Background] Shih YC, Chou CC, Lu YJ, Yu HY. Reliability and validity of the traditional Chinese version of the GAD-7 in Taiwanese patients with epilepsy. J Formos Med Assoc. 2022 Nov;121(11):2324-2330. doi: 10.1016/j.jfma.2022.04.018. Epub 2022 May 16. PMID 35584970
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Background] Krause SJ, Backonja MM. Development of a neuropathic pain questionnaire. Clin J Pain. 2003 Sep-Oct;19(5):306-14. doi: 10.1097/00002508-200309000-00004. PMID 12966256
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Leung GT, de Jong Gierveld J, Lam LC. Validation of the Chinese translation of the 6-item De Jong Gierveld Loneliness Scale in elderly Chinese. Int Psychogeriatr. 2008 Dec;20(6):1262-72. doi: 10.1017/S1041610208007552. Epub 2008 Jul 1. PMID 18590603
- [Background] Lee LL, Chiu YY, Ho CC, Wu SC, Watson R. The Chinese version of the Outcome Expectations for Exercise scale: validation study. Int J Nurs Stud. 2011 Jun;48(6):672-80. doi: 10.1016/j.ijnurstu.2010.11.001. Epub 2010 Dec 3. PMID 21129743
- [Background] Levis B, Sun Y, He C, Wu Y, Krishnan A, Bhandari PM, Neupane D, Imran M, Brehaut E, Negeri Z, Fischer FH, Benedetti A, Thombs BD; Depression Screening Data (DEPRESSD) PHQ Collaboration; Che L, Levis A, Riehm K, Saadat N, Azar M, Rice D, Boruff J, Kloda L, Cuijpers P, Gilbody S, Ioannidis J, McMillan D, Patten S, Shrier I, Ziegelstein R, Moore A, Akena D, Amtmann D, Arroll B, Ayalon L, Baradaran H, Beraldi A, Bernstein C, Bhana A, Bombardier C, Buji RI, Butterworth P, Carter G, Chagas M, Chan J, Chan LF, Chibanda D, Cholera R, Clover K, Conway A, Conwell Y, Daray F, de Man-van Ginkel J, Delgadillo J, Diez-Quevedo C, Fann J, Field S, Fisher J, Fung D, Garman E, Gelaye B, Gholizadeh L, Gibson L, Goodyear-Smith F, Green E, Greeno C, Hall B, Hampel P, Hantsoo L, Haroz E, Harter M, Hegerl U, Hides L, Hobfoll S, Honikman S, Hudson M, Hyphantis T, Inagaki M, Ismail K, Jeon HJ, Jette N, Khamseh M, Kiely K, Kohler S, Kohrt B, Kwan Y, Lamers F, Asuncion Lara M, Levin-Aspenson H, Lino V, Liu SI, Lotrakul M, Loureiro S, Lowe B, Luitel N, Lund C, Marrie RA, Marsh L, Marx B, McGuire A, Mohd Sidik S, Munhoz T, Muramatsu K, Nakku J, Navarrete L, Osorio F, Patel V, Pence B, Persoons P, Petersen I, Picardi A, Pugh S, Quinn T, Rancans E, Rathod S, Reuter K, Roch S, Rooney A, Rowe H, Santos I, Schram M, Shaaban J, Shinn E, Sidebottom A, Simning A, Spangenberg L, Stafford L, Sung S, Suzuki K, Swartz R, Tan PLL, Taylor-Rowan M, Tran T, Turner A, van der Feltz-Cornelis C, van Heyningen T, van Weert H, Wagner L, Li Wang J, White J, Winkley K, Wynter K, Yamada M, Zhi Zeng Q, Zhang Y. Accuracy of the PHQ-2 Alone and in Combination With the PHQ-9 for Screening to Detect Major Depression: Systematic Review and Meta-analysis. JAMA. 2020 Jun 9;323(22):2290-2300. doi: 10.1001/jama.2020.6504. PMID 32515813